CLINICAL TRIAL: NCT03483883
Title: A Phase I/IB Study of Avelumab in Combination With Gemcitabine for Advanced Renal Cell Carcinoma With Sarcomatoid Differentiation
Brief Title: Avelumab/Gemcitabine in Sarcomatoid RCC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to protracted accrual and limited patient engagement in the setting of rapidly changing treatment paradigms for advanced RCC with sarcomatoid features and/or intermediate/poor risk clinical features.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02818
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Metastatic sRCC
MeSH Terms: interventions — avelumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: Avelumab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Avelumab — Avelumab IV 10 mg/kg every 2 weeks
Drug: Gemcitabine — Dose Level 1: Gemcitabine 1250 mg/m2 IV every 2 weeks Dose Level 2: 1500 mg/m2 IV every 2 weeks

SUMMARY:
To determine the feasibility and safety of avelumab and gemcitabine combination therapy in patients with metastatic sRCC.

ELIGIBILITY:
Inclusion Criteria:

* Histologic evidence of metastatic RCC with sarcomatoid features (≥10% sarcomatoid component) or poor-risk RCC prognostic features (as defined by IMDC criteria). (14) An outside pathology report is sufficient for study eligibility. However, pathology should still be obtained as possible for internal institutional pathology review.
* ≥ 18 years of age.
* Phase I dose-escalation portion only:

Patients must have ≤3 prior systemic treatment regimens with recent evidence of disease progression by RECIST 1.1 criteria. Previous treatment with immune-checkpoint inhibitor therapy is allowable as a line of systemic therapy for the phase I portion. Prior systemic therapy in the adjuvant treatment setting is allowable as a prior line of therapy.

Phase Ib dose-expansion portion only:

Patients must have been treated with 0 or 1 prior lines of systemic therapy. Previous treatment with immune-checkpoint inhibitor therapy is allowable as a line of systemic therapy for the phase Ib expansion portion.

* No prior therapy with gemcitabine chemotherapy.
* ECOG performance status of 0-1. Patients must have primary or metastatic FFPE tissue available for histologic confirmation and possible determination of percent sarcomatoid component (if applicable).

Outside pathology report is sufficient for study eligibility. However, pathology should still be obtained as possible for internal institutional pathology review.

* Patients with history of treated brain metastases are eligible if off systemic corticosteroids for at least 2 weeks.
* Patients must have normal organ function, as confirmed by laboratory values obtained ≤ 14 days prior to the first day of study therapy:

Hematologic: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused) Hepatic: Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range and AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).

Renal: Estimated creatinine clearance ≥ 45 mL/min using Cockroft Gault formula.

* Patients must have a projected life expectancy of at least 3 months.
* PREGNANCY AND CONTRACEPTION:

Pregnancy test: Negative serum or urine pregnancy test at screening for women of childbearing potential.

Contraception: Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last avelumab treatment administration if the risk of conception exists.

In addition, women must not breastfeed while on this study as study drugs may also affect a breast-feeding child. Pregnant women and women who are breastfeeding are not allowed to participate in this study.

Exclusion Criteria:

* IMMUNOSUPRESSANTS: Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* AUTOIMMUNE DISEASE: Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* ORGAN TRANSPLANTATION: Prior organ transplantation including allogenic stem-cell transplantation.
* INFECTIONS: Active infection requiring systemic therapy.
* HIV/AIDS: Known history of testing positive for HIV or known acquired immunodeficiency syndrome, or positive HIV test result at screening.
* HEPATITIS: Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* VACCINATION: Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
* HYPERSENSITIIVTY TO STUDY DRUG: Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* CARDIOVASCULAR DISEASE: Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* OTHER PERSISTING TOXICITIES: Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Narayan, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States